CLINICAL TRIAL: NCT01771861
Title: Evaluation of a University Hospital Trauma Team Activation Protocol: a Prospective Cohort Study
Brief Title: Evaluation of Trauma Team Activation Criteria
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1912 (REK)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Trauma; Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Seriously injured or potentially seriously injured patients
  Interventions: Other: Trauma team activation

INTERVENTIONS:
Other: Trauma team activation — When admitting a potentially seriously injured patient, a trauma team is activated when prehospital information fulfills one or more prespecified criteria. The trauma team consist of a group of medical personnel including a surgeon, anesthesiologist and radiologist.

SUMMARY:
The aim of the study is to establish the predictive properties of our trauma team activation protocol, and its individual criteria, and if possible to suggest changes that reduce over- and undertriage.

The study will also give an overview of the frequency and type of emergency procedures at a university hospital trauma center, which can contribute to optimal resource use and indicate which type of surgical skills are necessary in our trauma emergency procedures.

DETAILED DESCRIPTION:
1. Background Multidisciplinary trauma teams reduce mortality and have become an important part of modern trauma care. Activation of the trauma team (TTA) when receiving patients with potentially severe injuries and protocols for TTA, are widely implemented throughout Scandinavia. Trauma team activation guidelines vary somewhat among Scandinavian trauma centers, but resemble the recommendations from the American College of Surgery - Committee On Trauma (ACS-COT). The criteria are based on parameters of physiologic compromise, anatomic injury classification, and mechanism of injury (MOI). They are designed to prevent undue delay of vital care as the trauma team is activated when prehospital information indicates that at least one of the TTA criteria is fulfilled. A substantial overtriage (activation of the trauma team despite only minor or moderate injury) is common and may reach 70%, mostly reflecting the limited precision of criteria relating to MOI. Overtriage is mainly a resource problem, as assembly of the multidisciplinary trauma team diverts personnel from other important activities in the hospital. Undertriage delays diagnosis and treatment of severely injured patients and may compromise the clinical outcome and even increase mortality. ACS-COT suggests that an overtriage as high as 50% is acceptable in order to minimize undertriage.

   Triage criteria should be adapted to the local case-load and injury pattern, which may vary considerably between geographical regions. The predictive properties of triage criteria depend on the prevalence of severe injuries. Typical for most Scandinavian trauma hospitals is a predominance of blunt over penetrating injuries. Furthermore, the frequency of severe polytrauma admissions is low.

   In 2011, we published an evaluation of the trauma team activation protocol in our hospital, leading to a change in the criteria. This study represents an evaluation of those changes and also addresses whether there may be a potential for further improvements.
2. Aim of the study The aim of the study is to establish the predictive properties of our TTA protocol, and its individual criteria, and if possible to suggest changes that reduce over- and undertriage.

   The study will also give an overview of the frequency and type of emergency procedures at a university hospital trauma center, which can contribute to optimal resource use and indicate which type of surgical skills are necessary in our trauma emergency procedures.
3. Method Identification of patients and inclusion-/exclusion criteria The trauma register at UNN Tromsø registers all patients admitted with TTA. Also included are patients with penetrating injury to the head/neck/torso/extremities proximal for elbow or knee, all patients with New Injury Severity Score (NISS) >12 and all patients with a head injury with AIS≥3. Excluded from the trauma register are patients with a chronic subdural hematoma, and patients with injuries from drowning, inhalation and asphyxia (strangulation/hanging).

   From the patients in the trauma register in the time period 1.2.2013 - 31.01.2015, we will identify and include patients.

   Data collection Almost all necessary data will be available from the trauma register. Criteria used for activation of the trauma team, is not registered in the trauma registry, and hence, will be registered from the documentation in the emergency medical dispatch centre (AMK) in Tromsø.

   Classification of injuries All injuries will be classified according to the Abbreviated Injury Scale (AIS)) and the extent of injuries will be classified with the Injury Severity Scale (ISS). Both classifications will be performed by authorized registrars.

   Triage The TTA protocol is evaluated against two standards, ISS and emergency procedure. Triage is considered correct when ISS>15 or an emergency procedure is performed aimed at stabilizing respiration or circulation. Overtriage is defined as the fraction of TTA where the patients are not severely injured (ISS≤15) or did not receive an emergency procedure. Undertriage is defined as the fraction of severely injured (ISS>15) or an emergency procedure was performed, and the patient was admitted without TTA.

   The ability of a criterion to predict severe trauma and/or need for an emergency procedure, is given as the percentage of patients that fulfilled the specific criterion that also had an ISS >15 and/or were subject to an emergency procedure.

   Hypothesis Previously, there was an undertriage of 12 % and an overtriage at UNN Tromsø of 70 %. On the 01.04.2011, the trauma team activation protocol at UNN Tromsø was revised, and of the previously 27 criteria, five criteria had been removed. We plan to assess if the current protocol has lead to an improvement in under- and overtriage. We also want to identify criteria which are seldom used (< 5 % of patients) and/or with a low positive predictive value (< 10 %), and these criteria will be considered omitted.

   A last hypothesis is to analyze if "walking wounded" is safe to admit without mobilizing the trauma team (a "walking wounded" patient is an injured patient with no loss of conscience and is up and walking on his own), given that there is enough prehospital information to assess this.
4. Design The study is a prospective cohort study, based on data from the trauma register at UNN Tromsø.
5. Parameters

   Baseline characteristics for included patients are:
   * sex
   * age
   * mechanism of injury
   * classification of injuries with AIS and ISS
   * transfer from other hospitals

   Outcome parameters include
   * type and frequency of emergency procedures performed at the local hospital and at UNN Tromsø
   * Criteria used for trauma team activation.
   * mortality

   Emergency procedures includes:
   * Chest tube insertion
   * Hemostatic surgery in the abdomen
   * Hemostatic surgery in the pelvis with packing
   * Thoracotomy
   * Primary stabilization of fractures (external fixation)
   * Endotracheal intubation (our addition)
6. Statistical methods Simple statistical methods like frequency, mean, median and percentage will be used.
7. Study group Supervisor is dr.med. Kristian Bartnes, Avd. for hjerte-/lunge-/karkirurgi, UNN.

   Coworkers are dr.med. Knut Fredriksen, Akuttmedisinsk avd. UNN; cand.med. Svein Arne Monsen, Anestesiavd. UNN and cand.med. Trond Dehli, Gastrokirurgisk avd, UNN.

   Trond Dehli is responsible for the practical follow-up of the study.
8. Time Schedule Data collection will start 1.2.13 and continue until 31.01.15. Since registration of data in the trauma registry most likely will be delayed by 2-12 weeks, the registration of data will continue until all patients in the registry are completed. Presentation of the study in the form abstract/posters and a manuscript will be written during 2015.
9. Ethics and publication The protocol will be sent to the regional ethical committee for approval. We plan to present the results in national and international conferences, and also in a peer-reviewed medical journal.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted with the trauma team
* all patients admitted with Injury Severity Score >15

Exclusion Criteria:

* secondary admittance(transfers)>24 post injury

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severly injured and potentially severly injured patients admitted at the University Hospital North Norway
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2013-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Trauma team activation criteria | 1 day
  The specific criterium or criteria that was fulfilled and was used to activate the trauma team

SECONDARY OUTCOMES:
Emergency procedure | 2 days
  All prespecified emergency procedures to stabilize airways, breathing and circulation will be registered.
Mortality | up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital North Norway, Tromsø, Norway